CLINICAL TRIAL: NCT04139902
Title: PHASE II NEOADJUVANT STUDY OF PD-1 INHIBITOR DOSTARLIMAB (TSR-042) VS. COMBINATION OF TIM-3 INHIBITOR COBOLIMAB (TSR-022) AND PD-1 INHIBITOR DOSTARLIMAB (TSR-042) IN RESECTABLE STAGE III OR OLIGOMETASTATIC STAGE IV MELANOMA (NEO-MEL-T)
Brief Title: Neoadjuvant PD-1 Inhibitor Dostarlimab (TSR-042) vs. Combination of Tim-3 Inhibitor Cobolimab (TSR-022) and PD-1 Inhibitor Dostarlimab (TSR-042) in Melanoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Diwakar Davar (Other)
Collaborators: Tesaro, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Diwakar Davar, Assistant Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 19-047
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Melanoma Stage III; Melanoma Stage IV
MeSH Terms: conditions — Melanoma | interventions — dostarlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dostarlimab (TSR-042) (singly) (Experimental): Pre-Operative Phase:
  Dostarlimab (TSR-042) 500mg will be administered through an IV over 30 minutes, on Cycle 1 Day 1, and then again on Cycle 2 Day 1.
  Post-Operative Phase:
  Dostarlimab (TSR-042) 500mg will be administered through an IV over 30 minutes for 4 doses every 3 weeks (Cycles 3-4) and then 1000mg will be administered through an IV over 30 minutes every 6 weeks for 6 doses (Cycles 5-10) for approximately 48 weeks.
  Interventions: Drug: Dostarlimab (TSR-042) (singly)
- Dostarlimab (TSR-042) and Cobolimab TSR-022 (combination) (Experimental): Pre-Operative Phase:
  Dostarlimab (TSR-042) 500mg and Cobolimab TSR-022 300mg will be administered through an IV over 30 minutes, on Cycle 1 Day 1 and then again on Cycle 2 Day 1.
  Post-Operative Phase:
  Dostarlimab (TSR-042) will be administered through an IV over 30 minutes for 4 doses every 3 weeks (Cycles 3-4), and then 1000mg will be administered through an IV over 30 minutes every 6 weeks for 6 doses (Cycles 5-10) for approximately 48 weeks. TSR-022 will not be administered.
  Interventions: Drug: Dostarlimab (TSR-042) and TSR-022 (combination)

INTERVENTIONS:
Drug: Dostarlimab (TSR-042) (singly) — If patients are randomized to Dostarlimab (TSR-042) alone, during the Pre-operative Phase, 500mg will be administered through an IV over 30 minutes, on Cycle 1 Day 1, and then again on Cycle 2 Day 1.
  Surgery will occur 1-4 weeks after completion of the pre-operative phase.
  During the Post-operative phase, Dostarlimab (TSR-042) 500mg will be administered through an IV over 30 minutes for 4 cycles every 3 weeks (Cycles 3-4), and then 1000mg will be administered through an IV over 30 minutes every 6 weeks (Cycles 5-10) for approximately 48 weeks.
  Other Names: Dostarlimab
  Arms: Dostarlimab (TSR-042) (singly)
Drug: Dostarlimab (TSR-042) and TSR-022 (combination) — If patients are randomized to the combination, Dostarlimab (TSR-042) and TSR-022, during the Pre-operative Phase, Dostarlimab (TSR-042) 500mg and TSR-022 300mg will be administered through an IV over 30 minutes on Cycle 1 Day 1 and then again on Cycle 2 Day 1.
  Surgery will occur 1-4 weeks after completion of the pre-operative phase.
  During the Post-operative Phase, Dostarlimab (TSR-042) 500mg will be administered through an IV over 30 minutes for 4 cycles every 3 weeks (Cycles 3-4) and then 1000mg will be administered through an IV over 30 minutes every 6 weeks for 6 doses (Cycles 5-10) for approximately 48 weeks.
  Arms: Dostarlimab (TSR-042) and Cobolimab TSR-022 (combination)

SUMMARY:
The purpose of this study is to test the effects of anti-PI-1 inhibitor (TSR-042) or anti-PD-1/anti-TIM-3 combination (TSR-042 / TSR-022) in patients with operable melanoma.

DETAILED DESCRIPTION:
This is a randomized phase II neoadjuvant study comparing neoadjuvant therapy with PD-1 inhibitor Dostarlimab (TSR-042) to the PD-1/TIM-3 inhibitor combination Dostarlimab (TSR-042)/TSR-022 in patients with resectable regionally advanced or oligometastatic melanoma.

Patients with stage III B/C/D or oligometastatic stage IV A melanoma with lymph node (LN) and/or in-transit and/or oligometastatic disease who have yet to undergo definitive surgery are eligible to enroll.

Suitable patients will be identified pre-operatively. Patients will undergo screening evaluation consisting of systemic/CNS staging scans, tumor biopsy, blood studies to confirm suitability. Subjects will receive neoadjuvant therapy (Dostarlimab (TSR-042) or Dostarlimab (TSR-042)/TSR-022 combination for 6 weeks prior to planned surgery (pre-operative phase). Surgery will occur 1-4 weeks after completion of pre-operative therapy. After recovery from surgery subjects will receive Dostarlimab (TSR-042) (Post-Operative phase) for approximately 48 weeks; for a total of 54 weeks of study drug(s) administration in total.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent for the study
* ≥ 18 years of age
* histologically or cytologically confirmed diagnosis of cutaneous or unknown primary melanoma (excluding uveal/choroidal and mucosal melanoma; although acral melanoma is included) belonging to one of the following AJCC 8th edition TNM stages:

  1. Tx or T1-4 AND
  2. N1b, or N1c, or N2b, or N2c, or N3b, or N3c AND/OR
  3. M1a or M1b

Patients are eligible for this trial either at presentation for primary melanoma with concurrent regional nodal and/or in-transit metastasis and/or oligometastasis; AND/OR at the time of clinical detected nodal and/or in-transit and/or oligometastatic recurrence; and may belong to any of the following groups:

Primary melanoma with clinically apparent regional lymph node metastases; Clinically detected recurrent melanoma at the proximal regional lymph node(s) basin; Clinically detected primary melanoma involving multiple regional nodal groups; Clinical detected nodal melanoma (if single site) arising from an unknown primary; In-transit and/or satellite metastases with or without regional lymph node involvement; Distant skin and/or in-transit and/or satellite metastases with or without regional lymph node involvement; Oligometastatic lung disease with or without regional lymph node involved permitted if deemed resectable at baseline NOTE: Determination of resectability must be made at baseline to be eligible for this neoadjuvant study.

* measurable disease based on RECIST 1.1
* must provide tumor tissue from a newly obtained core, punch, incisional or excisional tumor biopsy
* 0 or 1 on the ECOG Performance Scale
* Demonstrate adequate organ function on screening labs obtained within 14 days of registration
* negative serum pregnancy test (females of childbearing potential)
* females of non-childbearing potential must be ≥45 years of age and has not had menses for >1 year; if amenorrhoeic for <2 years without history of a hysterectomy and oophorectomy must have an FSH value in the postmenopausal range; post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation (documented hysterectomy or oophorectomy)
* male subjects should agree to use an adequate method of contraception

Exclusion Criteria:

* Patients with uveal and/or mucosal melanoma histology are excluded (Patients with melanoma of unknown histology are permitted to enroll after discussion with Principal Investigator)
* Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.
* Is receiving systemic immunosuppression with either corticosteroids (>10mg daily prednisone equivalent) or other immunosuppressive medications) for active autoimmune disease: history of active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids (>10mg daily prednisone or equivalent) or systemic immunosuppressive agents
* ≥ CTCAE grade 3 immune-related AE (irAE) experienced with prior immunotherapy (except, non-clinically significant lab abnormalities (elevations in lipase, amylase not associated with clinically significant disease etc.) even if ≥ CTCAE grade 3 may enroll if resolved at this time, or, development of autoimmune disorders of Grade ≤ 3 may enroll if the disorder has resolved to Grade ≤ 1)
* received prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent (except ≤ Grade 2 neuropathy)
* autoimmune disorders of Grade 4 while on prior immunotherapy
* active (i.e., symptomatic or growing) central nervous system (CNS) and/or leptomeningeal metastases (CNS lesions that are treated and deemed stable (repeat imaging study done at least 2 weeks prior to first dose of study treatment) are NOT permitted to enroll even if other inclusion criteria are met and patients are neurologically asymptomatic)
* known additional malignancy that is progressing or requires active treatment (except, basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy)
* invasive cancer diagnosed and treated less than 2 years prior to current presentation (other indolent malignancies that are not progressing and/or deemed to require active therapy are not exclusionary)
* evidence of interstitial lung disease or active, non-infectious pneumonitis
* active infection requiring systemic therapy
* history or current evidence of any condition, therapy, or laboratory abnormality determined to be significant, in the opinion of the treating investigator
* known psychiatric or substance abuse disorders that would interfere with study compliance
* is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial
* had a live vaccine within 30 days of initiating protocol therapy
* received prior therapy with an IDO inhibitor, anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137 and/or combination (including nivolumab, pembrolizumab or ipilimumab/nivolumab). Prior treatment with ipilimumab or interferon alfa is allowed.
* history of allergic or hypersensitivity reaction to components or excipients of Dostarlimab (TSR-042) and TSR-022, interferon alfa or ipilimumab
* known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* known history of or screening test that is positive for hepatitis B virus (HBV; eg, HBsAg reactive or HBV DNA detected) or hepatitis C virus (HCV; HCV antibody positive and/or HCV RNA quantitative is detected). Hepatitis C antibody - positive subjects who received and completed treatment for hepatitis C that was intended to eradicate the virus may participate if hepatitis C RNA levels are undetectable. Hepatitis B positive subjects who received and completed treatment for hepatitis B that was intended to eradicate the virus may participate if hepatitis B DNA levels are undetectable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2025-09-29 (Actual); Study Completion 2029-12-15 (Estimated)

PRIMARY OUTCOMES:
Major Pathologic Response (MPR) | 5 years (for population)
  Proportion of patients with an RVT (residual volume of viable tumor) of ≤10% remaining in post-therapy specimen using immunotherapy-specific pathologic assessment of neoadjuvant treated melanoma specimens.

SECONDARY OUTCOMES:
Number of Participants Experiencing Adverse Events Attributed to Treatment | Up to 56 months
  Number of participants experiencing adverse events (per CTCAE v5.0) that are possibly, probably or definitely related to study treatment, will be tabulated by category, grade and relatedness.
Frequency of Delays in Surgery | Up to 56 months
  Number of delayed of surgeries.
Frequency of Cancellations of Surgery | Up to 56 months
  Number of canceled surgeries.
Relapse-free Survival | Up to 56 months
  The length of time from initiation of study drug(s) until melanoma relapse (disease progression) as defined by RECIST v1.1, or death. Progressive Disease (PD): ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.
Overall Survival (OS) | Up to 56 months
  The length of time from initiation of study drug(s) that patients remain alive.

OTHER OUTCOMES:
Percentage of Circulating immune cells | Up to 56 months
  Percentage of immune cells present in circulating peripheral blood.
Percentage of Intratumoral immune cells | Up to 56 months
  Percentage of immune cells present in tumor.

CONTACTS AND LOCATIONS:
Overall Officials: Diwakar Davar, MD, Principal Investigator — UPMC Hillman Cancer Center
Locations (5):
- United States (5):
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center Washington, Washington, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gorry C, McCullagh L, O'Donnell H, Barrett S, Schmitz S, Barry M, Curtin K, Beausang E, Barry R, Coyne I. Neoadjuvant treatment for stage III and IV cutaneous melanoma. Cochrane Database Syst Rev. 2023 Jan 17;1(1):CD012974. doi: 10.1002/14651858.CD012974.pub2. PMID 36648215